#### **Title**

A Multicenter Randomized Placebo-Controlled Trial of Intravenous Thyroxine for Heart-Eligible Brain Dead Organ Donors

NCT: 04415658

**APPENDIX A: Study Forms** 

**Document Date: 01 December 2020** 

### A Multi-OPO Randomized Control Trial of T4 vs Placebo | Screening Worksheet #1

\*To be filled out on <u>EVERY</u> Brain-dead donor

| OPO: | |
|---|---|
| Donor UNOS #: | |
| Date: / | / 20 (mm/dd/yyyy) |
| <b>Inclusion Criteria</b> | : (Must have <u>ALL 4</u> inclusion criteria) |
| 1 | Declared dead by neurologic criteria |
| 2 | Authorization for organ donation <u>and</u> research |
| 3 | Donor age 14-55 years inclusive, <u>and</u> weight ≥ 45 kg (100 lbs.) |
| | Must be on 1 or more of the following vasopressors and/or inotropes at the start of ne study: |
| | <ul> <li>a norepinephrine</li> <li>b epinephrine</li> <li>c neosynephrine</li> <li>d dopamine</li> <li>e dobutamine</li> <li>f milrinone</li> </ul> |
| Exclusion Criteria | : (Must <u>NOT</u> have any exclusion criteria) |
| 2<br>3<br>4 | Brain-death declared >24 hours ago CAD or MI (by hx, EKG, or previous cardiac cath) that would exclude transplantation Significant valvular heart disease (by hx or echo) that would exclude transplantation Previous sternotomy or cardiac surgery |
| 6<br>7 | Donor is in a VA hospital Received IV or po T4/T3 in the last month (including home medication) Known HIV+ serology Other reason: |
| | has all 4 inclusion criteria and <u>no</u> exclusion criteria, he/she is eligible for the be randomized to either T4 or NS, and the infusion should be started as *** |
| ELI | GIBLE (go to worksheet) NOT ELIGIBLE – STOP! |

All worksheets are to be submitted to the OPO research coordinator

#### Worksheet #2

# Multi-OPO Randomized Control Trial of T4 vs Placebo Data Collection Worksheet UNOS number: (ravised 11/5/2020)

| OPO: | (revised 11/5/2020) |
|---|---|
| 1. Admission to the hospital: Date: / / 20; Time:: | (all times in 24:00) |
| 2. Brain Death: Date:/ / 20; Time: | : |
| Go to Sharepoint, Multi-OPO T4 RCT randomization sheet to identify the | next randomization |
| 3. Randomized to: T4 NS | |
| ***Draw <i>free T4, TSH</i> prior to starting T4 / NS infusion. | |
| 4a. Baseline results before starting T4 or saline: Weight kg | |
| 4b. Vent settings: f Vt cc FiO2 PEEP PaG | 02 |
| Labs: (most recent <u>before</u> starting protocol) [enter 999 if data not ava | ilable] |
| c. Highest Troponin I (before starting protocol) ng/ml d. ALT e. AST | |
| f. Bilirubin<br>g. Creatinine BUN | |
| h. Amylase | |
| i. INR<br>j. Calcium (total) <i>or</i> k. Calcium (ionized) | - |
| 5. T4 or NS started: Date: / / 20; Time:: | |
| (needs to be started within 24 hours of brain-death declaration) | |
| (needs to be started within 24 nours of brain-death declaration) | |
| 6. T4 rate: 30mcg/hr [ 500 mcg/ 500 cc NS at 30 cc/hr = 30 mcg/hr] a. Was T4 started at 30 mcg/hr Yes No | |
| b. If No, what was the reason: | |

| be | IS rate 30 cc/hr [should be equal to the normal T4 dose, i.e. 30 cc/hr] <i>The donor may</i> e on additional IV fluids as needed, but needs to have a separate IV of NS @ 30 cc/hr to natch the fluid intake with the T4 protocol. a. Was NS started at 30 cc/hr? Yes No b. If No, what was the reason: |
|---|---|
| *** | Please fill out the Multi-OPO RCT T4 Vasopressor Flow Sheet #3. |
| | only allowed doses of T4 are 30 mcg/hr, 20 mcg/hr, 10 mcg/hr. Decrease the dose by 'hr, if a lower dose is needed.*** |
| If<br>a.<br>b.<br>c. | Vas the T4 dose <u>decreased</u> before 12 hours? Yes No<br>Yes, what was the reason? (check all that apply) Tachycardia (HR increased more than 20 bpm over baseline and is > 120 bpm) Hypertension (Systolic BP increased >30 mmHg and is >180 mmHg) Arrhythmia: a fib/flutter; SVT; V tach; PVCs(>6/min) Other: |
| If<br>a.<br>b.<br>c. | Vas the T4 dose stopped before 12 hours? Yes No Yes, what was the reason? (check all that apply) Tachycardia (HR increased more than 20 bpm over baseline and is > 120 bpm) Hypertension (Systolic BP increased >30 mmHg and is >180 mmHg) Arrhythmia: a fib/flutter; SVT; V tach; PVCs(>6/min) Other: |
| Da | Time first echo <b>ordered</b> after T4/NS started: ate: / / 20; Time:: Ejection Fraction from first echo:% |
| 60 | f the donor was on T4 and completed the 12-hour protocol, was the T4 stopped within 0 minutes after the 12-hour study period? If the T4 stopped before 12 hours, answer /A and go to #15. Yes [skip to #15] No [go to #13] N/A [skip to #15] |

If the donor was in the NS group, skip to question #14.

| 13. What was the reason the T4 was continued beyond the study period? a. Still on vasopressors b. Still on inotropes c. Physician's preference d. Other e. Dose of T4 mcg/hr f. Time T4 stopped: Date: / / 20; Time:: Go to Question #15. |
|---|
| 14. If the donor was randomized to NS, did the donor receive T4 after enrollment in the study ("open-label")? Yes No |
| If yes, what was the reason? a. Still on vasopressors b. Still on inotropes c. Physician's preference d. Other |
| e. Dose of open-label T4 mcg/hr f. Time open-label T4 started: Date: / 20; Time:: g. Time open-label T4 stopped: Date: / 20; Time:: |
| 15. If more than 1 echo was performed, fill in the data below: [enter 999 in EF if not done] a. 2 <sup>nd</sup> echo: EF% Date://20; Time:: b. 3 <sup>rd</sup> echo: EF% Date://20; Time:: c. 4 <sup>th</sup> echo: EF% Date://20; Time:: |

## Draw *free T4* before going to the OR or at end of donor management on all donors in the study (T4 and control group)

| 16. <u>Baselin</u> | e Serum free T4 ng/dl | TSH mIU/I |
|---|---|---|
| 17. Serum | free T4 level ng/dl <u>prio</u> | r to OR. |
| 18.Was he | art transplanted ? Yes No _ | |
| a<br>b<br>c<br>d<br>e<br>f<br>j<br>k<br>l | not transplanted, what was the real Decreased EF, poor function, CAD: 1 vessel 2 vessel LVH Size Medical history (smoking, diabeted) Positive serologies Increased risk Match list exhausted Recipient issues Intra-op decline Surgical injury Valvular disease Other | 3 vessel |

| <b>ADVERSE EVENTS</b> : Please identify <b>any new</b> adverse events that occurred in the donor, <b>regardless if they received T4 or NS</b> , after the start of the study: |
|---|
| 19. Did the donor experience any of the following adverse events? Yes No If YES, please check all that occurred: |
| a Severe hypertension (BP >200 mm Hg) |
| b Tachycardia (HR> 150; including sinus tach, SVT, PSVT) |
| c Fever (>102 degree) |
| d A fib or a flutter |
| e Ventricular ectopy (>6 VPCs/min, bigeminy, trigeminy) |
| f V tach (spontaneously resolved) |
| g V tach (requiring cardioversion) |
| h V fib (requiring defibrillation) |
| i cardiac arrest* |
| j cardiac death prior to the OR* |
| k new skin rash |
| l other: |
| 19 m. Was the adverse event related to the T4 infusion? |
| YES NO UNCERTAIN |
| 19 n. Please describe the adverse event: |
| *These events need to be reported to the DSMB. |
| 20. Name of person filling out worksheet: |
| Date: |

**For the Research Coordinator:** After the case is completed, please upload the SRTR data to the Excel Spread sheet.

| T4 Vasopre | essor Flow | Sheet a | #3 | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| UNOS #: | | | OPO: | | Date Enrolled: | | [randomized to T4: or NS:] | | | | | | |
| | | BLOOD PRESSURE | | | | VASOPRESSOR AND INOTROPE DOSES (ENTER ZERO IF NOT ON THE DRUG) | | | | | | | |
| INTERVAL | Time<br>(Military)<br>(HR:min) | T4 Dose (mcg/ hr) | Saline<br>Dose<br>(cc/hr) | Heart<br>Rate | □ Invas | | Levophed*<br>(mcg/min) | Epi*<br>(mcg/kg/<br>min) | Neo*<br>(mcg/min) | Dopamine<br>(mcg/kg/<br>min) | Dobutrex*<br>(mcg/kg/<br>min) | Milrinone<br>(mcg/kg/<br>min) | Vaso*<br>(U/hr) |
| | | ''' ) | | | Sys | Dias | | | | | | | |
| BASELINE<br>Before first<br>dose of<br>T4/NS | ÷ | | | | | | | | | | | | |
| 2 HOURS | : | | | | | | | | | | | | |
| 4 HOURS | : | | | | | | | | | | | | |
| 6 HOURS | : | | | | | | | | | | | | |
| 8 HOURS | : | | | | | | | | | | | | |
| 10 HOURS | : | | | | | | | | | | | | |
| 12 HOURS | : | | | | | | | | | | | | |
| END OF<br>DONOR<br>MGMT <sup>1</sup> | | | | | | | | | | | | | |
| | | Date Va | asopressor<br>Ended | _/_/_ | // | // | // | _/_/_ | // | | | | |
| 12-hour output: ml | | | Time Va | asopressor<br>Ended | : | : | : | : | : | : | | | |
| 12-hour NE | | | | | | | *Norepinephrine | *Epinephrine | *Neosynephrine | | *Dobutamine | | *Vasopressin |
| Date/Time T | 4 stopped | (Use Mil | itary Tim | e): | | at | <b>:</b> | | | | | | |
| Notes/Comr | | | | | | | | | | | | | |
| Name of coo | prainator fil | iing out | worksne | eτ: | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> End of Donor Management is defined as when the donor was sent to the OR or was extubated in the ICU if no organs are procured.